CLINICAL TRIAL: NCT02597595
Title: Effects of Spirulina on Cardiac Functions in Children With Beta Thalassemia Major
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Professor Mohamed Elshanshory, professor and head of hematology and oncology unit at pediatric department, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2771/09/14
Record Dates: First submitted 2015-09-05; First posted 2015-11-05 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Beta Thalassemia
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patients (Experimental): thirty children with beta thalassemia major, with age range from 4-18 years, will receive oral spirulina (tablets=500 mg) for 3 months with a dose of 250 mg/kg/day (maximum dose 4 gm)
  Interventions: Other: spirulina
- controls (No Intervention): thirty healthy children of matched age and sex

INTERVENTIONS:
Other: spirulina — oral spirulina (tablet=500mg) will be given to patients for 3 months in a dose of 250 mg/kg/day (maximum 4 gm)
  Arms: patients

SUMMARY:
The aim of this study is to evaluate the cardioprotective effect of spirulina in children with beta thalassemia.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the cardioprotective effect of spirulina in children with beta thalassemia.

this study will be carried on thirty children with beta thalassemia major from those attending the Hematology Unit of Pediatric department at Tanta University Hospital, and another thirty healthy children of matched age and sex will be enrolled as controls.

all studied children will be subjected to careful history taking and through clinical examination. laboratory investigations will be done including complete blood count, hemoglobin electrophoresis, serum ferritin, liver and kidney functions, and troponin-1 plasma level. echocardiographic assessment of the cardiac functions will be done for all patients. Source data will be the patients medical records.

oral spirulina will be given for studied patients for 3 months, and clinical examination, laboratory investigations and cardiac functions will be assessed at the time of inclusion in the study, and again after 3 months of regular spirulina supplementation.

An informed consent will be obtained from parents of all included subjects. the results of this study will be tabulated and statistically analyzed using Statistical Package for the Social Sciences (SPSS).

ELIGIBILITY:
Inclusion Criteria:

* children suffering from beta thalassemia major with age range from 4-18 years

Exclusion Criteria:

* children with congenital heart diseases children with rheumatic heart diseases presence of heart failure children with coronary arterial disease children with cardiomyopathy

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
cardiac functions measured by echocardiography | after 3 months of regular oral spirulina supplementation
  Fractional shortening [FS]. Mitral flow early phase filling velocity [E], peak atrial phase filling velocity[A] and E/A ratio, and left ventricular (LV) diastolic function

SECONDARY OUTCOMES:
cardiac functions measured by troponin-1 plasma level. | after 3 months of regular oral spirulina supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Magda M Ibrahim, M.B.B.ch, Principal Investigator — Master Degree student; Osama AR Tolba, MD, Study Chair — supervisor; Rasha M Gamal, MD, Study Director — supervisor
Locations (1):
- Faculty of Medicine- Tanta University, Tanta, Gharbia Governorate, Egypt

REFERENCES:
- [Background] Khan M, Shobha JC, Mohan IK, Naidu MU, Sundaram C, Singh S, Kuppusamy P, Kutala VK. Protective effect of Spirulina against doxorubicin-induced cardiotoxicity. Phytother Res. 2005 Dec;19(12):1030-7. doi: 10.1002/ptr.1783. PMID 16372368
- [Background] Cogliandro T, Derchi G, Mancuso L, Mayer MC, Pannone B, Pepe A, Pili M, Bina P, Cianciulli P, De Sanctis V, Maggio A; Society for the Study of Thalassemia and Hemoglobinopathies (SoSTE). Guideline recommendations for heart complications in thalassemia major. J Cardiovasc Med (Hagerstown). 2008 May;9(5):515-25. doi: 10.2459/JCM.0b013e3282f20847. PMID 18404006
- [Background] Pennell DJ, Udelson JE, Arai AE, Bozkurt B, Cohen AR, Galanello R, Hoffman TM, Kiernan MS, Lerakis S, Piga A, Porter JB, Walker JM, Wood J; American Heart Association Committee on Heart Failure and Transplantation of the Council on Clinical Cardiology and Council on Cardiovascular Radiology and Imaging. Cardiovascular function and treatment in beta-thalassemia major: a consensus statement from the American Heart Association. Circulation. 2013 Jul 16;128(3):281-308. doi: 10.1161/CIR.0b013e31829b2be6. Epub 2013 Jun 17. PMID 23775258